CLINICAL TRIAL: NCT06670911
Title: A Phase II Trial of Low-dose Pembrolizumab Plus Chemotherapy for the First-Line Treatment of Persistent, Recurrent, or Metastatic Cervical Cancer - ACCESS I
Brief Title: Low-dose Pembrolizumab Plus Chemotherapy for the First-Line Treatment of Persistent, Recurrent, or Metastatic Cervical Cancer.
Acronym: ACCESS-I
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCESS-I
Record Dates: First submitted 2024-08-27; First posted 2024-11-01 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Persistent, Recurrent, or Metastatic Cervical Cancer
MeSH Terms: conditions — Recurrence | interventions — pembrolizumab; Drug Therapy; Paclitaxel; Carboplatin; Cisplatin

STUDY DESIGN:
Intervention Model Description: This is a phase II, Simon 2-stage study. The null hypothesis is that the response rate with chemotherapy alone is 0.35 (35% according to published data from the INCA (10)), and the alternative hypothesis is that the true response rate is 0.55 (20% increase in response with the addition of pembrolizumab, as per the KEYNOTE-826 study. In stage I, a total of 14 patients will be treated. If there are 5 or fewer responses among these 14 patients, the study will be terminated early. Otherwise, an additional 30 patients will be treated in stage II, resulting in a total sample size of 44. If there are 21 or more responses among these 44 patients, we reject the null hypothesis and conclude that the treatment is promising. The type I error is 0.05 and the power is 0.8.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low-dose Pembrolizumab Plus Chemotherapy (Experimental): pembrolizumab 100mg intravenous infusion plus chemotherapy every 3 weeks. Chemotherapy may consist of paclitaxel 175 mg/m² + carboplatina AUC 5 or paclitaxel 175 mg/m² + cisplatin 50 mg/m² for patients who have not been previously exposed to cisplatin.
  Interventions: Drug: Low-dose Pembrolizumab Plus Chemotherapy (Paclitaxel plus Carboplatin or Cisplatin)

INTERVENTIONS:
Drug: Low-dose Pembrolizumab Plus Chemotherapy (Paclitaxel plus Carboplatin or Cisplatin) — Patients will receive pembrolizumab 100mg IV every 3 weeks plus chemotherapy (paclitaxel 175 mg/m² + carboplatin AUC 5 or paclitaxel 175 mg/m² + cisplatin 50 mg/m² for cisplatin-naïve patients).

SUMMARY:
This is a phase II single-arm study of low-dose pembrolizumab (100mg, fixed-dose) plus chemotherapy in women aged 18 years or older with histologically confirmed persistent, recurrent, or metastatic cervical cancer who are ineligible for curative-intent treatment (surgery and/or radiation therapy) and who have not been previously treated with systemic chemotherapy, with the exception of chemotherapeutic agents used as radiosensitizers (cisplatin or carboplatin concurrent with radiation therapy).

DETAILED DESCRIPTION:
This is a phase II single-arm study of low-dose pembrolizumab plus chemotherapy in women aged 18 years or older with histologically confirmed persistent, recurrent, or metastatic cervical cancer who are ineligible for curative-intent treatment (surgery and/or radiation therapy) and who have not been previously treated with systemic chemotherapy, with the exception of chemotherapeutic agents used as radiosensitizers (cisplatin or carboplatin concurrent with radiation therapy).

Participants must have measurable disease as defined by RECIST 1.1, as assessed by the local investigator/radiologist, and must provide a tumor tissue sample no older than 4 years for PD-L1 expression status determination. PD-L1 expression will be analyzed using the 22C3 antibody (Dako®) and classified according to the Composite Positive Score (CPS).

Treatment will consist of pembrolizumab 100mg administered by intravenous infusion plus chemotherapy every 3 weeks. Chemotherapy may be paclitaxel 175 mg/m2 plus carboplatin AUC 5 or paclitaxel 175 mg/m2 plus cisplatin 50 mg/m2 for patients not previously exposed to cisplatin. Both carboplatin and cisplatin should be administered immediately after paclitaxel. All study treatments should be administered on Day 1 (D1) of each 3-week treatment cycle. All participants should receive premedication to prevent severe hypersensitivity reactions according to local practice. Premedication should be administered after the pembrolizumab infusion and before chemotherapy.

During the treatment period, participants will have routine clinical visits for treatment administration, safety and well-being monitoring, and assessment of disease status changes.

Primary safety assessments will include physical examinations, vital signs, electrocardiography (ECG), hematology and biochemistry tests, thyroid function tests, and urinalysis. At each visit, adverse events will be assessed and graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 1 5.0. Study treatment doses may be interrupted or reduced (applicable only to chemotherapy) or discontinued in case of severe adverse events.

Imaging assessments will include computed tomography (CT) of the chest and magnetic resonance imaging (MRI) of the abdomen and pelvis. The first study imaging assessment will be performed at 9 weeks (63 days ± 7 days) from the date of Cycle 1 (C1) Day 1 infusion. Subsequent imaging should be performed every 9 weeks (63 days ± 7 days) until Week 54 and every 12 weeks (84 days ± 7 days) thereafter. Other imaging exams such as bone scintigraphy or brain imaging should be performed as clinically indicated.

Participants may interrupt or discontinue pembrolizumab and continue in the study. Similarly, participants may interrupt or discontinue chemotherapy and continue treatment with pembrolizumab.

Participants will receive study treatments until disease progression as defined by RECIST 1.1, unacceptable toxicities, intercurrent illness that precludes continued treatment, investigator's decision to withdraw the participant from treatment, withdrawal of consent, or administrative reasons requiring treatment discontinuation.

Participants may receive up to 6 cycles of paclitaxel-platinum (carboplatin or cisplatin). Participants may receive a maximum of 35 administrations of pembrolizumab (approximately 2 years). In the case of complete response (CR), study treatment may be discontinued at the investigator's discretion after the CR has been confirmed by radiographic imaging and the participant has received at least 2 cycles of pembrolizumab and to have completed a minimum of 8 total treatment cycles (approximately 24 weeks).

Participants who discontinue study treatment for reasons other than radiographic disease progression will be followed until documented disease progression by RECIST 1.1 criteria, initiation of new anticancer therapy, withdrawal of consent, loss to follow-up, or death.

After discontinuation of study treatment, participants may initiate subsequent anticancer treatments at the discretion of the treating physician and in accordance with local standard of care.

After verification of disease progression by RECIST 1.1 and/or initiation of subsequent oncological treatment, all participants will be followed up for overall survival (by telephone contact or in-person visits to the center) until withdrawal of consent, loss to follow-up, death, or until the study is completed or terminated early, whichever occurs first.

Symptomatic improvement is a recognized clinical benefit. Participants will complete the EuroQol EQ-5D-5L, EORTC QLQ-C30, and EORTC QLQ-CX24 to assess quality of life.

The study will begin when the first participant signs the Informed Consent Form and will end when the last participant completes the final study-related call or visit, withdraws from the study, or is lost to follow-up (i.e., the participant cannot be contacted by the investigator).

ELIGIBILITY:
Inclusion Criteria:

1. ) Female participants aged 18 years and older
2. ) Patients with persistent, recurrent, or metastatic squamous cell, adenocarcinoma, or adenosquamous cervical cancer, with PD-L1 CPS ≥ 1 expression, who have not received prior chemotherapy and are ineligible for curative surgery and/ or radiotherapy. Prior chemotherapy used as a radiosensitizer and completed at least 2 weeks before the scheduled date for C1D1 with resolution of all treatment-related toxicities is allowed. Adverse events due to prior treatments must be resolved to ≤ grade 1 or the participant's baseline. Neuropathy ≤ grade 2 or alopecia of grade ≤ 2 are eligible.
3. ) Not pregnant or breastfeeding a ) Fertile-age women with the potential to become pregnant must agree to follow contraceptive guidance during treatment and for at least 120 days after the last dose of pembrolizumab and 210 days after the last dose of chemotherapy. Abstinence is acceptable if it is the participant's usual lifestyle and preferred contraception.
4. ) The participant (or legal representative, if applicable) must provide written informed consent for the study. The participant may also provide consent for future biomarker research. However, the participant may participate in the main study without participating in future biomarker research.
5. ) Have measurable disease according to RECIST 1.1 criteria, as assessed by the local investigator/radiologist. Lesions located in a previously irradiated area are considered measurable only if progression has been demonstrated.
6. ) Have an archived tumor tissue sample (recurrent or metastatic cervical cancer) no older than 4 years or provide a biopsy of a previously unirradiated tumor lesion for prospective PD-L1 status determination, since only participants with PD-L1 expression CPS ≥ 1 will be included in the study.
7. ) Performance Status/Eastern Cooperative Oncology Group (ECOG) of 0 to 1 within 7 days prior to C1D1
8. ) Have adequate organ function, as indicated by the following laboratory values within 7 days prior to C1D1: a ) Absolute neutrophil count (ANC) ≥ 1,500/mcL; b ) Platelets ≥ 100,000/mcL; c ) Hemoglobin ≥ 9.0 g/dL - The criterion must be met without erythropoietin dependence and without transfusion in the last 2 weeks prior to Cycle 1 Day 1; d ) Creatinine ≤ 1.5 x upper limit of normal or creatinine clearance ≥ 60 mL/min for participants with creatinine levels > 1.5 x upper limit of normal - creatinine clearance (CrCl) should be calculated according to institutional standard using the Cockcroft-Gault formula; d ) Total serum bilirubin ≤ 1.5 x upper limit of normal; e ) AST and ALT ≤ 2.5 x upper limit of normal or ≤ 5 x upper limit of normal for participants with hepatic metastases; f ) International Normalized Ratio (INR) or Prothrombin Time (PT), Activated Partial Thromboplastin Time (aPTT) or Partial Thromboplastin Time (PTT) ≤ 1.5 x upper limit of normal, unless the participant is receiving anticoagulant, provided that PT or aPTT is within the therapeutic range for the intended use of anticoagulants.

Exclusion Criteria:

1. ) Positive urine pregnancy test within 72 hours prior to C1D1. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required;
2. ) Presence of known active central nervous system metastases and/or carcinomatous meningitis. Participants with known brain metastases may be included provided that the brain metastases have been previously treated (except with chemotherapy) and are radiographically stable. To demonstrate radiographic stability of previously treated brain metastases, a minimum of two post-treatment brain imaging evaluations are required: 1) The first brain image should be acquired after completion of the treatment of brain metastases. 2) The second image should be obtained during screening (i.e., within 28 days prior to the scheduled C1D1 date) and >4 weeks after the prior post-treatment brain image.Known brain metastases are considered active if any of the following criteria apply: a ) The brain image obtained during screening shows progression of existing metastases or the appearance of new lesions compared to brain images taken at least 4 weeks earlier b ) The neurological symptoms attributed to brain metastases have not returned to baseline; c) Steroid doses exceeding 10 mg of prednisone daily (or equivalent) were used to treat symptoms related to brain metastases within 28 days prior to the scheduled C1D1 date.
3. ) Presence of other known malignancies within the past 3 years. Participants with basal cell carcinoma or squamous cell carcinoma of the skin who have undergone potentially curative therapy are not excluded.
4. ) Having a diagnosis of immunodeficiency or being on chronic systemic steroid therapy (at doses greater than 10 mg daily prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the scheduled C1D1 date.
5. ) Having an active autoimmune disease that has required systemic treatment within the past 2 years (i.e., with the use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency) is permitted.
6. ) History of non-infectious pneumonitis requiring steroid use.
7. ) Having an active infection requiring systemic therapy.
8. ) Having a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required.
9. ) Having a known history of hepatitis B (defined as positive hepatitis B surface antigen [HBsAg]) or known active hepatitis C virus (defined as detectable HCV RNA [qualitative]). No testing for hepatitis B and hepatitis C is required .
10. ) Having a known history of active tuberculosis.
11. ) Having received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent, or any other immune checkpoint inhibitor (CTLA-4, OX40, LAG3, etc.).
12. ) Having received prior systemic chemotherapy for the treatment of advanced cervical cancer (chemotherapy used as a radiosensitizer and completed at least 2 weeks prior to the scheduled start date of cycle 1, day 1).
13. ) Not having recovered adequately from toxicities and/or complications of major surgery prior to the scheduled start date of cycle 1, day 1.
14. ) Having received radiotherapy within 2 weeks prior to the scheduled start date of cycle 1, day 1.
15. ) Having received a live vaccine within 30 days prior to the scheduled start date of cycle 1, day 1 (measles, mumps, rubella, varicella/zoster, yellow fever, rabies, Bacillus Calmette-Guérin (BCG), typhoid fever vaccine, etc.). Seasonal influenza vaccines are permitted.
16. ) Having a contraindication or hypersensitivity to any component of carboplatin, paclitaxel, or cisplatin
17. ) Currently participating or has participated in a study of an investigational agent or used an experimental device within 4 weeks prior to the scheduled start date of cycle 1, day 1.
18. ) History of allogeneic solid organ/tissue transplantation.
19. ) Having a known psychiatric disorder or substance abuse that may interfere with the study requirements.
20. ) To have a history or current evidence of any condition, therapy, or laboratory abnormality that could confound the study results, interfere with participation, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by Investigator | Up to approximately 46 months
  Proportion of participants with complete or partial response per RECIST 1.1 as assessed by the investigator/radiologist patients with a confirmed complete or partial response by RECIST 1.1

SECONDARY OUTCOMES:
Duration of Response (DOR) Per RECIST 1.1 as Assessed by Investigator | Up to approximately 46 months
  For participants who demonstrate CR or PR, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death. The DOR per RECIST 1.1 as assessed by Investigator is presented.
  documented progression or death in the absence of disease progression
Number of Participants Who Experienced an Adverse Event (AE) | Up to approximately 46 months
  An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experienced an AE is presented.
Quality of life during treatment | Baseline (Cycle 1 Day 1: Predose) and up to approximately 46 months
  Assessment of Quality of Life Through Specific Questionnaires
PFS Per RECIST 1.1 as Assessed by Investigator in All Participants | Up to approximately 46 months
  PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥ 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 as assessed by Investigator for all randomized participants is presented
OS in All Participants | Up to approximately 46 months
  OS was defined as the time from randomization to death due to any cause. The OS for all randomized participants is presented.
Cost evaluation of adding pembrolizumab | Up to approximately 46 months
  To examine the direct cost consequences of incorporating pembrolizumab
Number of Participants Who Experienced a Serious AE (SAE) | Up to approximately 46 months
  An SAE was defined as any untoward medical occurrence that, at any dose: a.) Resulted in death; b.) Was life-threatening; c.) Required inpatient hospitalization or prolongation of existing hospitalization; d.) Resulted in persistent or significant disability/incapacity; e.) Was a congenital anomaly/birth defect; f.) Other important medical events; h.) Was a new cancer (that is not a condition of the study) or i.) Was associated with an overdose. The number of participants who experienced an SAE is presented.
Number of Participants Who Experienced an Immune-related AE (irAE) | Up to approximately 46 months
  AEs associated with pembrolizumab exposure may be a result of an immune response. These irAEs may occur shortly after the first dose or several months after the last dose of pembrolizumab treatment and may affect more than one body system simultaneously. For this study irAEs included, but were not limited to: -Pneumonitis; Diarrhea/Colitis; Aspartate transaminase (AST)/Alanine transaminase (ALT) elevation or Increased bilirubin; Type 1 diabetes mellitus or Hyperglycemia; Hypophysitis; Hyperthyroidism; Hypothyroidism; Nephritis and Renal dysfunction; and Myocarditis. The number of participants who experienced an irAE is presented.

CONTACTS AND LOCATIONS:
Overall Officials: Andreia c Melo, PhD, Principal Investigator — Instituto Nacional de Câncer José Gomes de Alencar da Silva - INCA
Locations (1):
- Instituto Nacional de Cancer, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] Cohen PA, Jhingran A, Oaknin A, Denny L. Cervical cancer. Lancet. 2019 Jan 12;393(10167):169-182. doi: 10.1016/S0140-6736(18)32470-X. PMID 30638582
- [Background] Kitagawa R, Katsumata N, Shibata T, Kamura T, Kasamatsu T, Nakanishi T, Nishimura S, Ushijima K, Takano M, Satoh T, Yoshikawa H. Paclitaxel Plus Carboplatin Versus Paclitaxel Plus Cisplatin in Metastatic or Recurrent Cervical Cancer: The Open-Label Randomized Phase III Trial JCOG0505. J Clin Oncol. 2015 Jul 1;33(19):2129-35. doi: 10.1200/JCO.2014.58.4391. Epub 2015 Mar 2. PMID 25732161
- [Background] Colombo N, Dubot C, Lorusso D, Caceres MV, Hasegawa K, Shapira-Frommer R, Tewari KS, Salman P, Hoyos Usta E, Yanez E, Gumus M, Olivera Hurtado de Mendoza M, Samouelian V, Castonguay V, Arkhipov A, Toker S, Li K, Keefe SM, Monk BJ; KEYNOTE-826 Investigators. Pembrolizumab for Persistent, Recurrent, or Metastatic Cervical Cancer. N Engl J Med. 2021 Nov 11;385(20):1856-1867. doi: 10.1056/NEJMoa2112435. Epub 2021 Sep 18. PMID 34534429
- [Background] Ribas A, Hamid O, Daud A, Hodi FS, Wolchok JD, Kefford R, Joshua AM, Patnaik A, Hwu WJ, Weber JS, Gangadhar TC, Hersey P, Dronca R, Joseph RW, Zarour H, Chmielowski B, Lawrence DP, Algazi A, Rizvi NA, Hoffner B, Mateus C, Gergich K, Lindia JA, Giannotti M, Li XN, Ebbinghaus S, Kang SP, Robert C. Association of Pembrolizumab With Tumor Response and Survival Among Patients With Advanced Melanoma. JAMA. 2016 Apr 19;315(15):1600-9. doi: 10.1001/jama.2016.4059. PMID 27092830
- [Background] Kang SP, Gergich K, Lubiniecki GM, de Alwis DP, Chen C, Tice MAB, Rubin EH. Pembrolizumab KEYNOTE-001: an adaptive study leading to accelerated approval for two indications and a companion diagnostic. Ann Oncol. 2017 Jun 1;28(6):1388-1398. doi: 10.1093/annonc/mdx076. No abstract available. PMID 30052728
- [Background] Low JL, Huang Y, Sooi K, Ang Y, Chan ZY, Spencer K, Jeyasekharan AD, Sundar R, Goh BC, Soo R, Yong WP. Low-dose pembrolizumab in the treatment of advanced non-small cell lung cancer. Int J Cancer. 2021 Jul 1;149(1):169-176. doi: 10.1002/ijc.33534. Epub 2021 Mar 6. PMID 33634869